CLINICAL TRIAL: NCT03626181
Title: Using Multiple Brain-based Biomarkers to Validate and Predict Response to Theta Burst Stimulation as a New Treatment for Major Depressive Disorder
Brief Title: Biomarkers of Theta Burst Stimulation in Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Rajamannar Ramasubbu, Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001858; RT # 10016954 (Other: University of Calgary)
Record Dates: First submitted 2018-07-04; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active TBS-DLPFC (Experimental): There is only one arm. All participants will receive Theta Burst Stimulation (transcranial magnetic stimulation) of the dorsolateral prefrontal cortex.
  Interventions: Device: Theta Burst Stimulation ( Transcranial Magnetic Stimulation)

INTERVENTIONS:
Device: Theta Burst Stimulation ( Transcranial Magnetic Stimulation) — Participants will receive bilateral TBS, 5 times daily (15 minutes between), over 5 consecutive days (25 sessions total). In each session they will receive intermittent TBS (iTBS) over left dorsolateral prefrontal cortex (DLPFC), followed by continuous TBS (cTBS) over right DLPFC. Stimulation sites will be targeted with the Localite neuronavigation system and Visor2 software, and according to Talairach coordinates in relation to individual MRIs. Intensity will be standardized at 120% of RMT.
  The MagPro stimulator will deliver iTBS over left DLPFC with 1620 pulses in 54 triplet bursts (5Hz) with train duration of 2 seconds, and intertrain interval of 8 seconds. cTBS over right DLPFC will consist of 1620 pulses in 54 triplet bursts, train duration of 2 seconds, with no intertrain interval.

SUMMARY:
This study investigates the brain-based biomarkers of treatment response to accelerated theta burst stimulation (aTBS) in patients with Major Depressive Disorder resistant to pharmacological treatment(MDD) in an open label design.

DETAILED DESCRIPTION:
Theta burst stimulation (TBS) is a newer form of rTMS which requires less stimulation time and produces longer lasting post-stimulation effects in the cerebral cortex (4). It has been shown to be effective in inducing synaptic plasticity and has similar or better efficacy in treating depression compared to rTMS (4).Newer accelerated TBS (aTBS) protocols that condense stimulation sessions down to several days rather than weeks have shown similar response rates when compared to prolonged TBS protocols, also with similar tolerability and safety. In order to develop aTBS as an effective treatment for MDD, future research should focus on identification of reliable predictors for better outcome to TBS. The main objectives were: 1) To directly compare multiple different brain-based measures (neuroimaging and electrophysiology) to identify which has the most power in accurately predicting response to TBS compared to sham. 2) To track both short and long-term longitudinal electrophysiological (EEG) changes related to the therapeutic effects of TBS.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must meet the DSM-5 diagnostic criteria for single-episode Major Depressive Disorder (MDD).
2. Participant must have failed to respond to >1 but <4 classes of oral antidepressant treatments in the current episode of depression.
3. Participant must have a HAMD total score of at least 18

Exclusion Criteria:

1. The participant's depressive symptoms have previously demonstrated nonresponse to:

   * An adequate course of rTMS/TBS over DLPFC in the current major depressive episode, defined as at least 3 weeks of treatment, 5 times weekly
   * An adequate course of treatment with electroconvulsive therapy (ECT) in the current major depressive episode, defined as at least 7 treatments with unilateral/bilateral ECT.
2. Participant has received vagal nerve stimulation (VNS) or has received deep brain stimulation (DBS) in the current episode of depression.
3. Participant has a current or prior DSM-5 diagnosis of Axis I comorbidities, including psychosis, bipolar disorder, obsessive compulsive disorder, based upon clinical assessment and confirmed by the MINI.
4. Participant has a current or prior DSM-5 diagnosis of Axis II comorbidities, including severe borderline personality disorders, antisocial, schizotypal, schizoid personality disorders based upon clinical assessment and confirmed by the MINI.
5. Participant has severe suicidal ideation/plan/ intent.
6. Participant has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria.
7. Participant has a current or past history of seizures and neurological problems, e.g. head injury, stroke, progressive neurological disorder and complicated and unstable medical disorders, e.g. cardiovascular-related conditions, diabetes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Change from baseline at 5 days of TBS treatment
  Clinician administered questionnaire to asses clinical improvement and classify response and remission

SECONDARY OUTCOMES:
1. Montgomery-Åsberg Depression Rating Scale (MADRS) | Change from baseline at 5 days of TBS treatment
  A ten item clinician administered questionnaire to measure the severity of depressive symptoms on a 0 to 6 severity scale with higher scores indicating more severe depressive symptoms. Cut-off points include: 0 to 6 - symptom absent, 7 to 19 - mild depression, 30 to 34 - moderate, 35 to 60 - severe depression.
2. Hamilton Anxiety rating Scale (HAM-A) | Change from baseline at 5 days of TBS treatment
  A rating scale to measure the severity of anxiety symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
2. Columbia Suicide Severity Rating Scale ( CSSRS) | Change from baseline at 5 days of TBS treatment
  A suicidal rating scale devised by researchers at Columbia University. The presence of suicidal ideation score ranges from 1-5 and the intensity of the suicidal ideation ranges from 0-25 with higher scores indicating higher levels of intensity.
MGH Rumination questionnaire | Change from baseline at 5 days of TBS treatment
  Self administered 9 items scale to measure the severity of rumination. Each item is measured from 0-4 with a total score range of 0-36. Higher scores indicate more severe rumination.
Snaith-Hamilton Pleasure scale-Clinician administered (SHAP-C) | Change from baseline at 5 days of TBS treatment
  This is to evaluate the ability to enjoy/experience pleasure. Each item can score 0 or 1 with a total score possibility of 0-14. Higher scores represent higher anhedonia and 3 or over is considered abnormal.
36 item short form survey (SF-36) | Change from baseline at 5 days of TBS treatment
  This is to evaluate physical and emotional health.
Global Assessment of Functioning (GAF) | Change from baseline at 5 days of TBS treatment
  This is to evaluate psychological, social and occupational functioning
Resting state functional connectivity-Functional magnetic resonance imaging (rsfMRI) | Pretreatment baseline
  Temporal correlation of brain signals as measured by BOLD signals
Magnetic resonance spectroscopy (MRS) | Pretreatment baseline
  To measure glutathione and glutamate concentration in DLPFC and ACC
Electroencephalogram | Change from baseline at 5 days of TBS treatment
  To measure neuronal oscillations

CONTACTS AND LOCATIONS:
Overall Officials: Rajamannar Ramasubbu, MD,FRCPC,MSc, Principal Investigator — University of Calgary, Department of Psychiatry
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Duprat R, Desmyter S, Rudi de R, van Heeringen K, Van den Abbeele D, Tandt H, Bakic J, Pourtois G, Dedoncker J, Vervaet M, Van Autreve S, Lemmens GM, Baeken C. Accelerated intermittent theta burst stimulation treatment in medication-resistant major depression: A fast road to remission? J Affect Disord. 2016 Aug;200:6-14. doi: 10.1016/j.jad.2016.04.015. Epub 2016 Apr 19. PMID 27107779
- [Result] Desmyter S, Duprat R, Baeken C, Van Autreve S, Audenaert K, van Heeringen K. Accelerated Intermittent Theta Burst Stimulation for Suicide Risk in Therapy-Resistant Depressed Patients: A Randomized, Sham-Controlled Trial. Front Hum Neurosci. 2016 Sep 27;10:480. doi: 10.3389/fnhum.2016.00480. eCollection 2016. PMID 27729854
- [Result] Fitzgerald PB, Hoy KE, Elliot D, Susan McQueen RN, Wambeek LE, Daskalakis ZJ. Accelerated repetitive transcranial magnetic stimulation in the treatment of depression. Neuropsychopharmacology. 2018 Jun;43(7):1565-1572. doi: 10.1038/s41386-018-0009-9. Epub 2018 Feb 5. PMID 29467437
- [Result] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Result] Li CT, Chen MH, Juan CH, Huang HH, Chen LF, Hsieh JC, Tu PC, Bai YM, Tsai SJ, Lee YC, Su TP. Efficacy of prefrontal theta-burst stimulation in refractory depression: a randomized sham-controlled study. Brain. 2014 Jul;137(Pt 7):2088-98. doi: 10.1093/brain/awu109. Epub 2014 May 10. PMID 24817188
- [Result] Oberman L, Edwards D, Eldaief M, Pascual-Leone A. Safety of theta burst transcranial magnetic stimulation: a systematic review of the literature. J Clin Neurophysiol. 2011 Feb;28(1):67-74. doi: 10.1097/WNP.0b013e318205135f. PMID 21221011
- [Result] Bakker N, Shahab S, Giacobbe P, Blumberger DM, Daskalakis ZJ, Kennedy SH, Downar J. rTMS of the dorsomedial prefrontal cortex for major depression: safety, tolerability, effectiveness, and outcome predictors for 10 Hz versus intermittent theta-burst stimulation. Brain Stimul. 2015 Mar-Apr;8(2):208-15. doi: 10.1016/j.brs.2014.11.002. Epub 2014 Nov 6. PMID 25465290
- [Result] Blumberger DM, Maller JJ, Thomson L, Mulsant BH, Rajji TK, Maher M, Brown PE, Downar J, Vila-Rodriguez F, Fitzgerald PB, Daskalakis ZJ. Unilateral and bilateral MRI-targeted repetitive transcranial magnetic stimulation for treatment-resistant depression: a randomized controlled study. J Psychiatry Neurosci. 2016 Jun;41(4):E58-66. doi: 10.1503/jpn.150265. PMID 27269205
- [Result] Brunoni AR, Chaimani A, Moffa AH, Razza LB, Gattaz WF, Daskalakis ZJ, Carvalho AF. Repetitive Transcranial Magnetic Stimulation for the Acute Treatment of Major Depressive Episodes: A Systematic Review With Network Meta-analysis. JAMA Psychiatry. 2017 Feb 1;74(2):143-152. doi: 10.1001/jamapsychiatry.2016.3644. PMID 28030740
- [Result] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537